CLINICAL TRIAL: NCT03735732
Title: Neuronal Correlates of Priming on Goal-directed and Cue-dependent Behavior
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Sabine Frank, Research Associate, University Hospital Tuebingen
Other Study IDs: PIT_brain
Record Dates: First submitted 2018-07-18; First posted 2018-11-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Functional Magnetic Resonance Imaging; Habits; Eating Behavior
MeSH Terms: conditions — Habits; Feeding Behavior | interventions — PRIME protocol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- weight status
- mindset
  Interventions: Behavioral: prime

INTERVENTIONS:
Behavioral: prime — groups be confronted with health or palatability aspects of food items
  Groups: mindset

SUMMARY:
The current proposal aims to investigate neuronal correlates of implicit and explicit priming paradigms for changing cue-dependent and goal-directed nutritional behavior.

DETAILED DESCRIPTION:
Food choice and intake is a daily and throughout normal subject. However, for more and more people eating habits and the question of food choice are of increasing interest and in several cases even a problem. The prevalence of obesity has tripled in the last decades and it is even spoken of an obesity epidemic. Life style interventions to lose weight often fail on the long run, also because people fall back into former unhealthy eating habits. Various factors influence our daily food choice, not all of which are apparent to ourselves. Thus, food choice might be goal-directed and therefore conscious and reflective, yet in other circumstances the choice to eat something specific might be based on cue dependent processes which are automatic and thus difficult to control. Since a change in eating-behavior and long-lasting weight loss is most problematic to achieve, the current proposal aims to investigate neuronal correlates of implicit and explicit priming paradigms for changing cue-dependent and goal-directed nutritional behavior.

ELIGIBILITY:
Inclusion Criteria:

* experimental: participants with obesity
* control: participants with normal-weight

Exclusion Criteria:

* currently dieting
* intolerance to provided food
* cognitive impairment
* contraindications for fMRI measurements

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy lean and obese volunteers
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in neuronal correlates | before and 5 minutes after visually presented food items
  Change of BOLD response measured by fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tübingen, Tübingen, Germany